CLINICAL TRIAL: NCT05486247
Title: Molecular Characterization of Gliomas Using a Broad NGS Panel
Brief Title: Molecular Characterization of Gliomas Using a Broad Next Generation Sequencing (NGS)Panel
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Principal Investigator, Rania Romanidou, Dr Ourania Romanidou, Hellenic Cooperative Oncology Group
Other Study IDs: NGSGLIOMA
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Malignant Glioma
Keywords: Molecular profile; Mutational status
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissue section
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gliomas are the most common malignant primary brain tumors with poor prognosis. The genotyping of tumors using NGS platforms enables the identification of genetic alterations that constitute diagnostic, prognostic and predictive biomarkers.Here in, we investigated the molecular profile of 32 tumor samples from 32 patients with high grade gliomas by implementing a broad 80-gene targeted NGS panel while reporting their clinicopathological characteristics and outcomes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of high grade glioma based on tissue biopsy

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of high grade glioma treated in 2 centers of the Hellenic Cooperative Oncology Group (HeCOG).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of genetic alterations in patients with high grade glioma using a 80 gene NGS panel | April 2019 - December 2021
  The prevalence of genetic alterations in patients with high grade glioma using a 80 gene NGS panel